CLINICAL TRIAL: NCT00577005
Title: Levetiracetam (Keppra) Treatment for Cocaine Dependence in Methadone-Maintained Patients
Brief Title: Efficacy of Levetiracetam in Cocaine-Abusing Methadone Maintained Patients
Acronym: Keppra-DB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0707002832; 5R01DA017782-04 (NIH); NIDA-5R01DA017782-04; Yale-0508000534; VA-gg0006
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Cocaine Dependence; Opioid Dependency
Keywords: GABAergic; levetiracetam
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Levetiracetam tablets
  Interventions: Drug: levetiracetam
- 2 (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: levetiracetam — The participants will start receiving Levetiracetam 500mg in the mornings of the first day on week 2. The dose will be titrated every third day, until the target dose of 3000mg/day is achieved by week 4. The study medication must be titrated to 3000 mg/day or to the subject's maximum tolerated dose (MTD). The physician overseeing this titration as well as all study staff will be blind to the subject's medication administration. The medication will be discontinued over a two-week period.
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
Concurrent dependence on cocaine occurs in up to 50% of the over one million opiate dependent patients in spite of methadone maintenance treatment being highly effective for opiate dependence and having excellent treatment retention. Cocaine dependence has remained largely unresponsive to medications both in and outside of these methadone programs. We have initial data from our open-label study with levetiracetam showing that this medication is well tolerated and may reduce cocaine use in this cocaine-abusing methadone treated population.

The specific aim of this study is to evaluate the efficacy of levetiracetam 3 grams/day in modifying cocaine-using behavior, reducing cocaine craving and attenuating cocaine's reinforcing effect among methadone-maintained patients. The primary outcomes will be reduction in cocaine use as assessed by self-report and thrice-weekly urinalyses. Secondary outcomes will include weeks in treatment (retention) and change in measures of cocaine craving, anxiety symptoms and opiate withdrawal symptoms.

DETAILED DESCRIPTION:
This 17-week double-blind, placebo controlled randomized pilot clinical trial will provide treatment for 40 cocaine-dependent opioid dependent patients. Participants, aged 18-65 years, will be randomized to receive levetiracetam 3000 mg/day or placebo while concurrently receiving treatment with methadone. Baseline cocaine use will be determined during the first week of treatment participation. (Gossop et al., 1997) The study design will have three overlapping phases that are summarized below: 1) A one week methadone fixed induction (week 1) and flexible methadone stabilization phase (weeks 2-13); 2) an 12-week "treatment" phase (weeks 2-13), consisting of slow titration and stabilization on study medication; and 3) a four week "taper, detoxification or transfer" phase (weeks 13-17).

During the first week of induction onto methadone, participants will be administered increasing doses of methadone starting at 30 mg daily and increased up to 60 mg daily by the end of the first week. This methadone dose will be adjusted for stabilization of opiate withdrawal symptoms using a flexible dosing from 40 mg up to 150 mg between weeks 2 to 12. This range has been found to be adequate for the vast majority of patients receiving methadone in our program and is designed to accommodate participants who may not be able to tolerate the higher maintenance doses or may still experience withdrawal symptoms, respectively. We may increase or decrease this amount on a case-by-case basis based on physician assessment of self-reported and observed symptoms.

Starting on week 2 subjects will start study medication in one of two randomly assigned experimental groups: levetiracetam 3000 mg /day (active medication) or placebo (inactive medication). Concurrent with the stabilization on methadone, levetiracetam will be increased from 500mg/day on week 2 and this dose will be slowly titrated to a total of 3000mg/day or maximum tolerated dose (MTD). Subjects will remain on their full dosage through week 13.

At the end of week 13, participants will undergo detoxification from methadone over a 4-week period (weeks 13-17) and discontinuation from levetiracetam over a concurrent 2-week period.

All participants will receive weekly 1-hour of individual psychotherapy (Cognitive Behavioral Treatment) with experienced clinicians specifically trained to deliver the therapy and who will receive ongoing supervision. The primary outcomes will be reduction in cocaine use, as assessed by self-report and thrice-weekly urinalyses. Secondary outcomes will include weeks in treatment (retention), reported medication side effects (medication tolerability), and change in measures of: cocaine craving, anxiety symptoms and opiate withdrawal symptoms. This study will occur at the Outpatient Treatment Research Program in Building 36 at the VA CT Healthcare System.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65 years.
* Participants must demonstrate current opioid dependence as determined by study physician or APRN, self-reported history of opioid dependence for one year and a positive urine of opiates. Participants may be transferred from other methadone maintenance programs, including the WHVA methadone program.
* Participants also must be current users of cocaine with self-reported use of cocaine > 1 time/week in at least one month preceding study entry, cocaine-positive urine screen and score over 3 as assessed with the Severity Dependence Scale.
* Women of childbearing age are eligible to be included in the study if they have a negative pregnancy test at screening, agree to adequate contraception to prevent pregnancy, to have monthly pregnancy tests, and they understand the risk of fetal toxicity due to medication and cocaine.

Exclusion Criteria:

* Current diagnosis of other drug or alcohol dependence (other than opiates, cocaine or tobacco).
* Patients with serious medical illness (e.g., major cardiovascular, renal, endocrine, hepatic, and serious neurological disorders including any history of seizures).
* Patients with current serious psychiatric illness or history of psychosis, schizophrenia, bipolar type I disorder and subjects with suicidal or homicidal thoughts or taking psychotropic medications.
* Women who are pregnant, nursing or refuse to use a reliable form of birth control or refuse monthly testing.
* Screening liver function tests (SGOT or SGPT) greater than 3 times normal and renal function test (creatinine) greater than 1.5 mg/dl.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-07; Primary Completion 2008-06 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Gonzalez, MD, Principal Investigator — Yale University
Locations (1):
- VA CT Healthcare System, West Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty three cocaine and opioid dependent treatment seeking individuals were recruited by newspaper advertising, word-of -mouth and referrals from community-based substance abuse clinics. Research staff obtained informed consent and subjects were evaluated for study eligibility.
Pre-assignment Details: Twenty eight subjects were assigned to treatment groups while concurrently receiving treatment with methadone. Randomization was balanced with urn procedure on gender and severity of cocaine use score.
Groups:
- Levetiracetam 3000mg + Methadone: Participants were inducted onto methadone during the first week of study participation and then started on Levetiracetam 500mg in the mornings of the first day of week 2. The dose was titrated every third day on a twice day schedule, until the target dose of 3000mg/day was achieved or to the subject's maximum tolerated dose (MTD) by week 4.
  Levetiracetam: 3000mg orally everyday for 12 weeks
- Levetiracetam 0mg + Methadone: Participants were inducted onto methadone during the first week of study participation. Matching placebo capsules were started on week 2. The placebo capsules were given on a twice a day schedule until week 13.
  Placebo: Placebo orally everyday for 13 weeks
Period: Overall Study
Arm/Group | Levetiracetam 3000mg + Methadone | Levetiracetam 0mg + Methadone
Started | 16 | 12
Completed | 11 | 9
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Levetiracetam: Levetiracetam tablets
  levetiracetam: The participants will start receiving Levetiracetam 500mg in the mornings of the first day on week 2. The dose will be titrated every third day, until the target dose of 3000mg/day is achieved by week 4. The study medication must be titrated to 3000 mg/day or to the subject's maximum tolerated dose (MTD). The physician overseeing this titration as well as all study staff will be blind to the subject's medication administration. The medication will be discontinued over a two-week period.
- Placebo: matching placebo
  Placebo
- Total: Total of all reporting groups
Arm/Group | Levetiracetam | Placebo | Total
Number analyzed (Participants) | 16 | 12 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (10.7) | 33.6 (9.6) | 34.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 9 | 7 | 16
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 15 | 11 | 26
  African American | 0 | 1 | 1
  Hispanic | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change of Thrice Weekly Cocaine Free Urine Toxicology From Week 1 to 13
Description: The primary outcome variable was the change from baseline to week 13 of the thrice weekly cocaine-free urine scores. In this repeated ordinal variable, 0 represented all 3 urine samples submitted by the subject as positives, 1 represented some urine samples submitted by the subject were negative, and 2 represented all 3 urine samples submitted by the subjects were negative for cocaine. Balancing the distribution between these categories improved the models for the analysis of repeated ordinal data. Data is summarized as number of participant that were cocaine free urine (score 2) per week by group.
Time Frame: Weekly from baseline to week 12
Population: The intent-to-treat (ITT) sample were the 28 subjects were randomized and received one dose of study medication.
Measure: Number; unit: participants that were cocaine free
Arm/Group | Levetiracetam 3000mg + Methadone | Levetiracetam 0mg + Methadone
Number analyzed (Participants) | 16 | 12
participants that were cocaine free
  Baseline | 6 | 0
  week 1 | 3 | 2
  week 2 | 6 | 3
  week 3 | 5 | 4
  week 4 | 5 | 4
  week 5 | 5 | 2
  week 6 | 3 | 4
  week 7 | 3 | 3
  week 8 | 4 | 3
  week 9 | 4 | 4
  week 10 | 5 | 4
  week 11 | 5 | 5
  week 12 | 5 | 5
Statistical Analysis 1: Comparison: Levetiracetam 3000mg + Methadone vs Levetiracetam 0mg + Methadone; Test type: Superiority or Other; p = 0.09, Mixed Models Analysis — p-value <0.05 considered statistically significant; We modeled the the change in thrice weekly cocaine urines using a mixed-effect ordinal regression approach with MIXOR; Slope = -0.05425, Standard Error of Mean 0.03211 — Group x time interaction: Z=-1.68950 p = 0.09112

2. Secondary Outcome: Change of Thrice Weekly Opioid Free Urine Toxicology From Week 1 to 13
Description: The secondary outcome variable was the change from baseline to week 13 of the thrice weekly opioid-free urine scores. In this repeated ordinal variable, 0 represented all 3 urines samples submitted by the subject as positives, 1 represented some urine samples submitted by the subject were negative, and 2 represented all 3 urines samples submitted by the subjects were negative for opioids excluding methadone. Balancing the distribution between these categories improved the models for the analysis of repeated ordinal data. Data summarized by number of participants who were had opioid free urine samples (score 2) per week by group.
Time Frame: Weekly from baseline to week 12
Population: The intent-to-treat (ITT) sample were the 28 subjects were randomized and received one dose of study medication.
Measure: Number; unit: participants with opioid free urine
Groups:
- Levetiracetam 3000mg + Methadone: Participants were inducted onto methadone during the first week of study participation and then started on Levetiracetam 500mg in the mornings of the first day of week 2. The dose was titrated every third day on a twice day schedule, until the target dose of 3000mg/day was achieved or to the subject's maximum tolerated dose (MTD) by week 4.
  Levetiracetam: 3000mg orally everyday for 12 weeks
  .
Arm/Group | Levetiracetam 3000mg + Methadone | Levetiracetam 0mg + Methadone
Number analyzed (Participants) | 16 | 12
participants with opioid free urine
  Baseline | 4 | 4
  week 1 | 5 | 3
  week 2 | 7 | 4
  week 3 | 5 | 6
  week 4 | 6 | 3
  week 5 | 8 | 4
  week 6 | 7 | 4
  week 7 | 5 | 6
  week 8 | 5 | 4
  week 9 | 6 | 4
  week 10 | 6 | 5
  week 11 | 8 | 5
  week 12 | 5 | 5
Statistical Analysis 1: Comparison: Levetiracetam 3000mg + Methadone vs Levetiracetam 0mg + Methadone; Test type: Superiority or Other; p = 0.55, Mixed Models Analysis — p-value <0.05 considered statistically significant; We modeled the the change in thrice weekly opioid urines using a mixed-effect ordinal regression approach with MIXOR; Slope = 0.02570, Standard Error of Mean 0.04369 — Group x time interaction: Z= 0.58823 p = 0.55638

3. Secondary Outcome: Treatment Retention
Description: Weekly from week 1 to 13
Time Frame: Week 13
Population: Intent-treat-sample (ITT) that was inducted onto methadone and received one dose of study medication on week 2.
Measure: Number; unit: participants
Arm/Group | Levetiracetam 3000mg + Methadone | Levetiracetam 0mg + Methadone
Number analyzed (Participants) | 16 | 12
participants | 13 | 9
Statistical Analysis 1: Comparison: Levetiracetam 3000mg + Methadone vs Levetiracetam 0mg + Methadone; Test type: Superiority or Other; p = 0.67, Log Rank — p-value <0.05 considered statistically significant; Chi-Square 0.175. df = 1, p=0.676

4. Secondary Outcome: Cocaine Craving
Description: Weekly cocaine craving was measure at intake and weekly after with the Visual Analog Scale (VAS) of the Cocaine Selective Severity Assessment. The VAS measures the intensity of cocaine craving with a scale from 0 (No desire at all) to 7 (Unable to resist), and frequency of cocaine craving in the previous 24 hours with a scale from 0 ( never) to 7 ( all the time). The scale is totaled for a maximum number of 14, the minimum is 0. (Kampman et al., 1998; Mulvaney et al., 1999).
Time Frame: Weekly from baseline to week 12
Population: Intent to treat sample
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Levetiracetam | Placebo
Number analyzed (Participants) | 16 | 12
units on a scale
  Baseline | 7.19 (1.512) | 6.50 (1.617)
  week 1 | 4.13 (1.373) | 5.75 (1.488)
  week 2 | 2.64 (1.097) | 2.83 (1.192)
  week 3 | 2.13 (1.041) | 3.42 (1.417)
  week 4 | 2.13 (0.985) | 3.17 (1.140)
  week 5 | 2.53 (0.904) | 3.27 (1.556)
  week 6 | 3.00 (1.144) | 2.18 (1.278)
  week 7 | 2.67 (1.484) | 3.18 (1.470)
  week 8 | 2.80 (1.340) | 3.60 (1.454)
  week 9 | 2.33 (1.124) | 3.09 (1.486)
  week 10 | 2.18 (1.306) | 3.55 (1.603)
  week 11 | 2.09 (1.031) | 4.20 (1.800)
  week 12 | 3.27 (1.579) | 4.22 (1.985)
Statistical Analysis 1: Comparison: Levetiracetam vs Placebo; Test type: Superiority or Other; p = 0.11, Mixed Models Analysis — Significant p-value < 0.05; Slope = -0.1557 — Interaction of time x group: Z = -1.5671, p = 0.11708

ADVERSE EVENTS:
Time Frame: Adverse events were collected from week 1 to week 13
Arm/Group | Levetiracetam 3000mg + Methadone | Levetiracetam 0mg + Methadone
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 1/16 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam 3000mg + Methadone (N=16) | Levetiracetam 0mg + Methadone (N=12)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 2 (2)
Cut finger-accident (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes